CLINICAL TRIAL: NCT02990975
Title: Effect of Ultrasonography Guided Transversus Abdominis Plane Block to Intraoperative Anesthesia in Children: Randomized Controlled Study
Brief Title: Transversus Abdominis Plane Block In Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ERZINCAN UNIVERSITY 7
Record Dates: First submitted 2016-12-04; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Intra-operative Anesthesia
Keywords: Intra-operative anesthesia; Pediatric patient; Transversus Abdominis Plane Block
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- block and ketamine (Active Comparator): Transversus Abdominis Plane block after ketamine atropine induction and continued with ketamine only in anesthesia
  Interventions: Drug: ketamine
- ketamine atropine; laryngeal mask (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane MAC and oxygen / air mixture and applied Transversus Abdominis Plane block.
  Interventions: Drug: ketamine
- control group (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane MAC and oxygen / air mixture and Non-block, postoperative analgesia with paracetamol IV
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
Aim of this study; Intra-operative anesthesia and analgesia effects of Transversus Abdominis Plane Block supported by ketamine sedation only.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* To undergo elective lower abdominal surgery
* between 2-6 years old

Exclusion Criteria:

* Patients with psychiatric disease
* Patients whose weight is more than 40 kg
* Patients with cardiac-pulmonary-neurological disease
* Patients with bleeding disorder
* Patients with infection or scar on the injection area
* Patients with known allergies to local anesthetics

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the amount of anesthetic drug which was used | two hour

SECONDARY OUTCOMES:
Postoperative visual analogue scale | one day

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacroix F. Epidemiology and morbidity of regional anaesthesia in children. Curr Opin Anaesthesiol. 2008 Jun;21(3):345-9. doi: 10.1097/ACO.0b013e3282ffabc5. PMID 18458552
- [Background] Willschke H, Marhofer P, Machata AM, Lonnqvist PA. Current trends in paediatric regional anaesthesia. Anaesthesia. 2010 Apr;65 Suppl 1:97-104. doi: 10.1111/j.1365-2044.2010.06242.x. PMID 20377551
- [Background] Mishriky BM, George RB, Habib AS. Transversus abdominis plane block for analgesia after Cesarean delivery: a systematic review and meta-analysis. Can J Anaesth. 2012 Aug;59(8):766-78. doi: 10.1007/s12630-012-9729-1. Epub 2012 May 24. PMID 22622954
- [Background] Schaeffer E, Millot I, Landy C, Nadaud J, Favier JC, Plancade D. Another use of continuous transversus abdominis plane (TAP) block in trauma patient: pelvic ring fractures. Pain Med. 2014 Jan;15(1):166-7. doi: 10.1111/pme.12029. Epub 2013 Jan 7. No abstract available. PMID 23294595
- [Background] Niraj G, Kelkar A, Fox AJ. Application of the transversus abdominis plane block in the intensive care unit. Anaesth Intensive Care. 2009 Jul;37(4):650-2. doi: 10.1177/0310057X0903700420. PMID 19681428
- [Background] Walter CJ, Maxwell-Armstrong C, Pinkney TD, Conaghan PJ, Bedforth N, Gornall CB, Acheson AG. A randomised controlled trial of the efficacy of ultrasound-guided transversus abdominis plane (TAP) block in laparoscopic colorectal surgery. Surg Endosc. 2013 Jul;27(7):2366-72. doi: 10.1007/s00464-013-2791-0. Epub 2013 Feb 7. PMID 23389068
- [Background] Stuart-Smith K. Hemiarthroplasty performed under transversus abdominis plane block in a patient with severe cardiorespiratory disease. Anaesthesia. 2013 Apr;68(4):417-20. doi: 10.1111/anae.12108. Epub 2012 Dec 17. PMID 23252578
- [Background] Tekelioglu UY, Demirhan A, Sit M, Kurt AD, Bilgi M, Kocoglu H. Colostomy with Transversus Abdominis Plane Block. Turk J Anaesthesiol Reanim. 2015 Dec;43(6):424-6. doi: 10.5152/TJAR.2015.89410. Epub 2015 Dec 1. PMID 27366540